CLINICAL TRIAL: NCT04545697
Title: mHealth ElectroNic COnsultation REcording (mENCORE) in Advanced Prostate Cancer: a Feasibility Trial of a Patient Decision Support Intervention
Brief Title: mHealth ElectroNic COnsultation REcording (mENCORE) in Advanced Prostate Cancer
Acronym: mENCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20554; NCI-2020-07023 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Prostate Cancer
Keywords: Shared decision-making; Consultation audio recordings; Mobile health; mHealth
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Decision Support (Experimental): Instructions will be provided for installation and use of a smartphone recording app 7-60 days before an oncology consultation. Participants will share the recording with the Patient Support Corps (PSC), who will summarize the recording, send it to the participant's oncologist for review, then return an annotated summary to the participant within a week of the consultation.
  Interventions: Other: Medcorder

INTERVENTIONS:
Other: Medcorder — Medcorder is a smartphone app that is HIPAA compliant for the use of on patient recordings of consults with healthcare providers.

SUMMARY:
Patients surviving with advanced prostate cancer frequently encounter time points in their disease course that require choosing among multiple options regarding systemic therapy. Interventions to improve shared decision-making through patient support measures such as question listing, and audio recording and summarizing of consultations have been shown to improve patient-reported measures of decision making quality, e.g. decreased decisional conflict and regret. However, the feasibility of consultation recording and summarizing with mobile health (mHealth) technology on patient-owned smartphones is unknown. The investigators will conduct a single-arm trial to determine feasibility and acceptability of a clinician-prompted, patient administered smartphone audio recording application and a service to summarize the recordings (Patient Support Corps or PSC), in improving decision-making quality among patients with chemotherapy-naive, progressive, metastatic castration-resistant prostate cancer (mCRPC). This trial will inform the design and conduct of a larger trial evaluating broader scale implementation of this intervention.

DETAILED DESCRIPTION:
The intervention (provision of instructions on how to install/use the app and how to share the recording with the PSC) will take place 7-60 days before the upcoming oncology consultation. PSC will provide a summary within a week of the consultation.

Primary Objective:

To determine the percentage of enrolled participants who use a clinician-prompted, patient-administered smartphone application to create an audio recording of an outpatient oncology visit.

Secondary Objectives:

1. To determine the percentage of enrolled participants who listen to the audio recording within 1 week after the visit.
2. To determine the percentage of enrolled participants who request and receive a written summary of the consultation from the Patient Support Corps within 1 week after the visit.
3. To determine whether audio recording and summarization change decision-making quality measures.
4. To determine whether audio recording and summarization change provider-reported workload and other outcomes.
5. To determine whether audio recording and summarization change the frequency of follow-up communication between participant and clinic staff.

Participants will be followed via electronic medical record review for 2 weeks after consultation

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer of any histology.
2. Metastatic castrate-resistant Prostate Cancer (mCRPC)
3. Progression per any Prostate Cancer Working Group 3(PCWG3) criterion.
4. Has never received chemotherapy
5. Currently receiving or has previously received any androgen-signaling inhibitors (ASI) (abiraterone, enzalutamide, apalutamide, or darolutamide) that was discontinued due to progression
6. 18 years of age or older.
7. Able to read, speak, and write in English.
8. Has an upcoming genitourinary (GU) medical oncology appointment (in-person or Zoom video visit) at University of California, San Francisco (UCSF) within 7-60 days of enrollment.
9. Has access to and ability to use an iPhone (iOS) or Android smartphone.
10. Patient's UCSF oncology provider agrees to be recorded.

Exclusion Criteria:

1. Lack of decision-making capacity to provide consent to this trial.
2. Uncorrectable hearing or visual impairment hindering the ability to perform necessary tasks in the trial.
3. Any neurocognitive or psychiatric disorder hindering the ability to perform necessary tasks in the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of enrolled participants who utilized the application | Up to 2 weeks after the appointment
  Proportion of enrolled participants who create a complete audio consultation recording of the appointment using the application, measured by application metrics, at 1 week post-consultation along with 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Proportion of enrolled participants who listened to audio recording within 1 week after the visit | Up to 2 weeks after the appointment
  Proportion of enrolled participants who listen to the recording, measured by participant-reported survey at 1 week post-consultation along with 95% confidence interval will be reported.
Proportion of enrolled participants who obtain written summary of the consultation | Up to 2 weeks after the appointment
  Proportion of enrolled participants who request and receive a written summary of the consultation from the Patient Support Corps (PSC) within 1 week after the visit along with 95% confidence interval will be reported.
Mean participant-reported CollaboRATE scores | Up to 2 weeks after the appointment
  The CollaboRATE is a 3-item questionnaire developed to measure shared decision making in reference to the most recent appointment the participant may have had with the oncologist.
  The questions are as follows: (i) How much effort was made to help you understand your health issues? (ii) How much effort was made to listen to what matters most to you about your health is-sues? (iii) How much effort was made to include what matters most to you in choosing what to do next? Each response ranges from a score of 0-9, with a response of 0 = "No effort was made" and 9="Every effort was made". Higher total scores represent more shared decision making.
Mean score of participant reported Decision Regret Scale (DRS) | Up to 2 weeks after the appointment
  The DRS is a 5-item questionnaire where participants are asked to reflect on a past decision, and then asked to indicated the extent to which they agree or disagree with the statement in the regret scale by indication a number from 1 (Strongly) to 5 (Strongly Disagree) that best indicated their level of agreement. Scores are converted to a 0-100 scale with a lower scores indicating less regret.
Mean change in scores on the Informed subscale of the Decisional Conflict Scale (DCS) from baseline | Baseline and up to 2 weeks after the appointment
  The "Informed" subscale of the DCS consists of 3 items which measure the degree that the participant feel informed, with scores that range from 0 (strongly agree) to 4 (Strongly disagree). Scores are summed and then converted to a scale of 0-100, with lower indicating a greater degree of feeling informed. For analyzing changes in DCS information subscale, a two-tailed paired sample t-test will be used to determine whether the mean difference between pre- and post-consultation survey scores is 0 or not.
Mean perceived change in work burden provider-reported workload and other outcomes | Up to 2 weeks after the appointment
  The change in work burden will be determined using a provider-reported workload survey to determine whether audio recording produced a change in work burden at 1 week post-consultation among providers with enrolled participants. There are 5 possible responses: "Decreased work", "No Change", "A little more work", "Some more work", and "A lot more work".
Mean perceived change in provider-patient relationship quality | Up to 2 weeks after the appointment
  The change in provider-patient relationship quality will be determined using a provider-reported survey to determine whether audio recording produced a change in the provider patient relationship at 1 week post-consultation among providers with enrolled participants. There are 5 possible responses: "Negatively", "Somewhat Negatively", "No change", "Somewhat Positively", and "Positively".
Mean change in number of participant-initiated telephone call or portal message encounters over time | Baseline and up to 2 weeks after the appointment
  Changes in the frequency of follow-up communication between participant and clinic staff in the electronic health record from baseline (2 weeks pre-consultation to consultation) to post-consultation (consultation to 2 weeks post-consultation).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kwon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No